CLINICAL TRIAL: NCT06912763
Title: Reversing External-beam Radiotherapy-associated Fibrosis Syndrome: an Interventional Bayesian Adaptive Randomized-controlled Orphan Drug Platform Trial for Orodental Sequelae (Reverse-fibrose)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-1521; NCI-2025-02225 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Fibrosis Syndrome; Lymphedema; Head &Amp; Neck Cancer; Fibrosis
MeSH Terms: conditions — Lymphedema; Head and Neck Neoplasms; Fibrosis | interventions — Pravastatin; Pharmaceutical Preparations; Pentoxifylline; Ketoprofen; Standard of Care; Tocopherols

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment with Pravastatin QD (Experimental): 40 mg/day for 12 months
  Interventions: Drug: Pravastatin (drug)
- Treatment with Pentoxifylline TID + Tocopherol (Experimental): 400 mg/1000 IU vitamin E for 12 months
  Interventions: Drug: Pentoxifylline; Drug: tocopherol
- Treatment with Ketoprofen TID (Experimental): 75 mg for 12 months
  Interventions: Drug: ketoprofen
- Treatment with Pirfenidone TID (Experimental): 801 mg for 12 months
  Interventions: Drug: Pirfenidoneone
- Treatment with SoC (Control) (Experimental): No pharmacologic intervention (control)
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Drug: Pravastatin (drug) — Given PO
  Arms: Treatment with Pravastatin QD
Drug: Pentoxifylline — Given PO
  Arms: Treatment with Pentoxifylline TID + Tocopherol
Drug: ketoprofen — Given PO
  Arms: Treatment with Ketoprofen TID
Drug: Pirfenidoneone — Given PO
  Arms: Treatment with Pirfenidone TID
Other: Standard of Care (SOC) — SOC
  Arms: Treatment with SoC (Control)
Drug: tocopherol — Given PO
  Arms: Treatment with Pentoxifylline TID + Tocopherol

SUMMARY:
To find out if adding medication can help treat or prevent lymphedema and/or fibrosis related to radiation therapy, in survivors of head and neck cancer. Researchers will compare these drugs to find the most effective therapy for preventing or limiting these side effects.

DETAILED DESCRIPTION:
Primary Objectives

1. Determine the relative utility of candidate agents to reduce clinician-rated radiation lymphedema/fibrosis

   1. Hyp 1: Participants receiving candidate agent(s) will exhibit a proportional lower rate of Common Toxicity Criteria- Adverse Event (CTC-AE v5.0) rating of Grade 2 or greater on either "Fibrosis deep connective tissue" or "Superficial soft tissue fibrosis" by formal clinician assessment at 12 months post-randomization.
   2. Hyp 2: Participants receiving candidate agent(s) will exhibit a proportional lower rate of objective lymphedema/fibrosis rated as "moderate/severe" grade at any head and neck subsite as measured by the Head and Neck External Lymphedema and Fibrosis (HN-ELAF) Assessment Criteria by a certified lymphedema specialist at 12 months post-randomization.
2. Determine the relative effect size observed of candidate agent(s) to reduce objective imaging-derived measures of radiation lymphedema/fibrosis-related sequalae [Primary]

   1. Hyp 3: Participants receiving candidate agent(s) will exhibit a proportionally lower rate of objective DIGEST-detected swallowing dysfunction 12 months post-randomization.
   2. Hyp 4: Participants receiving candidate agent(s) will exhibit a proportional lower rate of objective MRI-detected difference between 6- and 18-month post-randomization quantitative T1 (T1 mapping) intensity for paired muscle swallowing/neck/masticator muscles receiving >=40Gy post-randomization.

Secondary Objectives

1. Determine the relative effect size observed of candidate agent(s) to reduce patient reported measures of toxicity associated with lymphedema/fibrosis-related sequalae [Secondary]

   1. Hyp 5: Participants receiving candidate agent(s) will exhibit a proportionally lower rate of moderate-severe rated items "Fibrosis deep connective tissue" or "Superficial soft tissue fibrosis" by patient self-assessment using the Participant Reported Outcomes-CTCAE (PROCTCAE) Scale at 12-months post-randomization.
   2. Hyp 6: Participants receiving candidate agent(s) will exhibit a proportionally lower rate of moderate-severe rated symptom items by participant self-assessment using the Head and Neck External Lymphedema and Fibrosis (HN-ELAF) Symptom Inventory Scale at 12-months post-randomization.
   3. Hyp 7: Participants receiving candidate agent(s) will exhibit a proportionally lower rate of moderate-severe global symptom burden by participant self-assessment using the MD Anderson Symptom Inventory Scale at 12-months post-randomization.
   4. Hyp 8: Participants receiving candidate agent(s) will exhibit a proportionally improved global quality of life as denoted by patient self-assessment using the EQ-5D Visual analogue Scale at 12-months post-randomization.

      .

ELIGIBILITY:
Eligibility Criteria Eligibility criteria (observational registry or randomization)

1. Prior history of head and neck cancer with no active disease.
2. Treated previously with radiotherapy with prescribed dose (greater or equal to 30Gy) to unilateral or bilateral neck(s)
3. Detectable CTC-AE G2+ lymphedema/fibrosis at >6 months post-radiotherapy.
4. No active liver disease (Child-Pugh class B-C), cirrhosis, nor active alcoholism, nor history of ulcers.
5. No history of myopathy/rhabdomyolysis.
6. Creatinine clearance <30mL/min.
7. No history of acute myocardial infarction or severe coronary disease.
8. Non-pregnant/post-menopausal, or male.
9. No history of diabetes mellitus
10. Allergy/hypersensitivity to HMG Co-A reductase inhibitor and/or xanthine derivatives, e.g., caffeine, theophylline, theobromine
11. No contraindications for magnetic resonance imaging a Subject to the discretion of the treating physician and Principal Investigator (PI), as the MRI may be optional

Exclusion Criteria

1. Active liver disease (Child-Pugh class B-C), cirrhosis, nor active alcoholism.
2. History of myopathy/rhabdomyolysis.
3. History of acute myocardial infarction or severe coronary disease.
4. Pregnant/post-menopausal, or male.
5. History of diabetes mellitus.
6. Allergy/hypersensitivity to Hydroxymethylglutaryl-coenzyme A (HMG Co-A) reductase inhibitor and/or xanthine derivatives, e.g., caffeine, theophylline, theobromine.
7. Contraindications for MRI Subject to the discretion of the treating physician and Principal Investigator (PI), as the MRI may be optional
8. Participants who are receiving any other investigational agents.
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition to statins, hemorheologic agents or other agents used in study
10. Participants with psychiatric illness/social situations that would limit compliance with study requirements.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2033-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events | Through study completion; an average of 1 year
  Incidence of Adverse of Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Clifton Fuller, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org